CLINICAL TRIAL: NCT03136614
Title: Prognostic Value of the Arteriograph in the Surgical Theatre and at the Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Zsolt Molnár, MD, PhD, DEAA, clinician, Szeged University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Arteriograph-2016
Record Dates: First submitted 2017-02-20; First posted 2017-05-02 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Anaesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Preoperative (Active Comparator): A single measurement with an Arteriograph is performed a day before an elective surgical intervention.
  Interventions: Device: Arteriograph
- Intraoperative (Active Comparator): An arteriograph is put on the patient for the time of operation. The device is set to measure in every 5 minutes.
  Interventions: Device: Arteriograph
- Intensive Care Unit (Active Comparator): Three separate measurements are performed on the subject with an Arteriograph throughout every dayshift for 3 days.
  Interventions: Device: Arteriograph

INTERVENTIONS:
Device: Arteriograph

SUMMARY:
To investigate how pulse wave velocity, aortic augmentation index and the arterial pulse wave given by the Arteriograph contributes to preoperative assesment, intraoperative and intensive care monitoring.

ELIGIBILITY:
Inclusion Criteria:

For the "preoperative" arm:

* Signed informed consent form
* Arterial catheter for hemodynamic monitoring

For the "intraoperative" arm:

* Signed informed consent form
* Arterial catheter for hemodynamic monitoring
* The operation will presumably last for more than 2 hours

For the "intensive care unit" arm:

* Signed informed consent form
* PiCCO monitor for hemodynamic monitoring

Exclusion Criteria:

For the "preoperative" arm:

* Pregnancy
* Subject belongs to a vulnerable group (ISO 14155:2011) e.g.: study member, medical student

For the "intraoperative" arm:

* Pregnancy
* Subject belongs to a vulnerable group (ISO 14155:2011) e.g.: study member, medical student
* Measuring blood pressure on both arms is not possible
* Insertion of an arterial catheter is not necessary or contraindicated
* Insertion of a central venous catheter is not necessary or contraindicated

For the "intensive care unit" arm:

* Pregnancy
* Subject belongs to a vulnerable group (ISO 14155:2011) e.g.: study member, medical student

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number and degree of hypotensive episodes predicted by preoperative values of pulse wave velocity. | One year
  The investigators will examine if high values of pulse wave velocity correlate with the frequency and severity of hypotensive episodes under anaesthesia.
Correlation between systemic vascular resistance and aortic augmentation index | One year
Identity of cardiac output given by the PiCCO monitor and cardiac output given by the Arteriograph | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Intensive Therapy, Szeged, Csongrád megye, Hungary

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — http://www.tensiomed.com/en/